CLINICAL TRIAL: NCT03318484
Title: Sonodynamic Therapy Manipulate Atherosclerosis Regression Trial Among Patients With Femoropopliteal PAD and Claudication
Brief Title: Sonodynamic Therapy on Patients With Femoropopliteal PAD and Claudication
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Re-registered
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Collaborators: Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ye Tian
Record Dates: First submitted 2017-10-12; First posted 2017-10-24 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2017-10

CONDITIONS: Peripheral Arterial Disease; Atherosclerosis; Cardiovascular Diseases
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal Medical Care (Active Comparator): Optimal medical care (OMC) only is administrated in this arm. OMC is established according to the standards established by the 2016 ACC-AHA Guidelines for the Management of Patients with Peripheral Artery Disease in order to promote best practices for risk factor management.
  Interventions: Drug: Optimal Medical Care
- Optimal Medical Care and SDT (Experimental): OMC and sonodynamic therapy (SDT) are administrated in this arm.
  Interventions: Drug: Optimal Medical Care; Combination Product: Sonodynamic therapy

INTERVENTIONS:
Drug: Optimal Medical Care — Aspirin 100mg once a day, Atorvastatin 20mg once a day and Antihypertensive Agents if necessary.
Combination Product: Sonodynamic therapy — SDT treatment is the combination of sonosensitizer administration and target atherosclerotic lesions ultrasound exposure. Sinoporphyrin sodium (DVDMS) as sonosensitizer, is dissolved in 0.9% sodium solution for following skin test and intravenous injection. 0.01mg/ml DVDMS solution (0.1ml) is prepared for skin test followed by 0.04 mg/ml DVDMS solution intravenous injection (0.2mg/kg). The target atherosclerotic lesions are marked on the corresponding skin with ultrasound guidance and underwent ultrasound exposure after 4 hours incubation. The therapeutic ultrasonic transducer is fixed to the marked skin site for 15min of each lesion. Ultrasound parameters included intensity of 1.8W/cm2 for femoral lesions, resonance frequency: 1.0 MHz and duty factor: 30%.
  Arms: Optimal Medical Care and SDT

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of sonodynamic therapy (SDT) in reducing atherosclerotic plaques inflammation and increasing peak walking time (PWT) among peripheral artery disease (PAD) patients with symptom of intermittent claudication.

DETAILED DESCRIPTION:
Atherosclerotic lower extremity PAD affects more than 20 million people in the world. PAD is associated with a major decline in functional status and claudication is the most frequent symptom. Current claudication therapies are associated with significant limitations. Pharmacotherapy cilostazol and supervised exercise are recommended in 2016 AHA/ACC Guideline on the management of lower extremity PAD patients with claudication, but cilostazol may not achieve an ideal response rate, and supervised exercise efficacy may be limited by co-morbidities and medicare reimburse. Furthermore endovascular procedure may not be feasible, durable or cost-effective, especially in femoropopliteal arteries.

The aim of this trial is to test the hypothesis that SDT improves PWT by inhibiting atherosclerotic plaques inflammation in femoropopliteal arteries PAD patients compared to optimal medical care (OMC) within 6 month. An estimated 80 eligible patients will be randomly divided into tow groups: OMC and SDT combined with OMC. Recruitment will be performed over 6 months and patients will be followed for 6 months; the anticipated total study duration will be 2 years.

Finally, this trial investigate the safety and efficacy of SDT in PAD patients with intermittent claudication and explore new end-points to evaluate therapeutic effects using PET-CT imaging as well as traditional endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with atherosclerotic peripheral artery disease with symptoms of moderate to severe intermittent claudication (defined as ability to walk at least 2, but not more than 11, minutes on a graded treadmill test using the Gardner protocol)
2. Aged ≥40 years
3. Resting ABI < 0.9 or ABI decreases > 0.15 after treadmill test regardless of the ABI at rest
4. Presence of significant stenosis but not occlusion of femoropopliteal arteries including the common femoral artery, superficial femoral artery and popliteal artery as determined by: Duplex ultrasound imaging OR lower extremity computed Tomography Angiography (CTA) OR lower extremity magnetic resonance angiography (MRA) OR lower extremity catheter-based contrast arteriography. Each of these noninvasive and invasive anatomic assessments will identify patients with at least a 50% stenosis in the affected segment
5. Stable use of low to moderate dose statin and the permitted statin drugs/doses: atorvastatin 20 mg, simvastatin 40 mg, rosuvastatin 10 mg, pravastatin, 40 mg, fluvastatin 80 mg or lovastatin 40 mg for at least 6 weeks prior to screening
6. Written informed consent

Exclusion Criteria:

1. Critical limb ischemia or other comorbid conditions that limit walking ability (claudication must be the consistent primary exercise limitation)
2. Inability to complete treadmill testing per protocol requirements
3. Two treadmill tests are completed at baseline to confirm reproducibility of results; those who deviates >25% are excluded
4. Severe aorto-iliac arteries stenosis or occlusion documented by noninvasive and invasive anatomic assessments
5. Allergic to DVDMS
6. Diagnosis of porphyria
7. Pregnant women and nursing mothers
8. Contraindications of PET/CT
9. Concurrent enrollment in another clinical trial
10. Presence of any clinical condition that in the opinion of the principal Investigator or the sponsor makes the patient not suitable to participate in the trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
PWT change, mins | Measured at baseline, 1, 3 and 6 months.
  Change from baseline peak walking time (PWT) at 6 months is assessed by graded treadmill test (Gardner protocol). The patient continues the test until walking can no longer be tolerated because of claudication symptoms.
MDS TBR change, (%) | Measured at baseline, 1 and 3 months.
  Change from baseline most disease segments (MDS) at 3 months is assessed by 18FDG-PET imaging. Uptake of FDG by the common and superficial femoral artery is expressed as the target, vessel wall to background, lumen ratio (TBR). The mean max MDS TBR is defined as the arterial segment centered on the slice of artery demonstrating the highest FDG uptake at baseline within the index vessel, and calculated as a mean of maximum TBR values derived from three contiguous axial segments.

SECONDARY OUTCOMES:
COT change, mins | Measured at baseline, 1, 3, and 6 months.
  Change from baseline claudication onset time (COT) at 6 months is assessed by graded treadmill test (Gardner protocol). The patient continues the test until calf muscle discomfort is first noticed.
AS TBR change, (%) | Measured at baseline, 1 and 3 months.
  Change from baseline active slice (AS) at 3 months is assessed by 18FDG-PET imaging. Uptake of FDG by the common and superficial femoral artery is expressed as the target, vessel wall to background, lumen ratio (TBR). The mean max AS TBR is defined as average mean maximal TBR of only slices with TBR >1.6 from index vessel at baseline.
WV TBR change, (%) | Measured at baseline, 1 and 3 months.
  Change from baseline whole vessel (WV) TBR at 3 months is assessed by 18FDG-PET imaging. Uptake of FDG by the common and superficial femoral artery is expressed as the target, vessel wall to background, lumen ratio (TBR). The mean max WV TBR is defined as a single whole vessel average mean maximal TBR of all the slices that compose the index vessel.
Serum inflammation cytokine level | Measured at baseline, 1, 3, and 6 months.
  Including Interleukin-6, Interleukin-1β, and high-sensitivity C-reactive protein (hs-CRP) level in serum
Pre-exercise ABI | Measured at baseline, 1, 3, and 6 months.
  Ankle-Brachial Index (ABI) is the ratio of the blood pressure at the ankle to the blood pressure of the upper arm. Pre-exercise ABI is collected routinely with the patient supine immediately prior to a treadmill test.
Post-exercise ABI | Measured at baseline, 1, 3, and 6 months.
  Ankle-Brachial Index (ABI) is the ratio of the blood pressure at the ankle to the blood pressure of the upper arm. Post-exercise ABI is collected routinely with the patient supine immediately following a treadmill test.
Intimal-medial thickness, (mm) | Measured at baseline, 1, 3, and 6 months.
  Estimation of the intimal-medial thickness for common femoral artery by doppler ultrasound.
Peak flow velocity, (cm/s) | Measured at baseline, 1, 3, and 6 months.
  Estimation of the systolic and diastolic peak flow velocity of the affected segments by doppler ultrasound.
Vessels' diameter, (mm) | Measured at baseline, 1, 3, and 6 months.
  Estimation of the vessels' diameter for common femoral artery by doppler ultrasound.
Diameter stenosis, (%) | Measured at baseline, 1, 3, and 6 months.
  Estimation of the maximum diameter stenosis of the affected segments by doppler ultrasound.
WIQ score | Measured at baseline, 1, 3, and 6 months.
  The Walking Impairment Questionnaire (WIQ) assesses the severity of the subjective walking impairment on distance, speed, and stair climbing scales. It is administered as a self report. Range: Minimum score is 0.2, maximum 100.
SF-36 score | Measured at baseline, 1, 3, and 6 months
  The patient reported SF-36 data assesses subjective physical limitations, leg symptoms, social function, treatment satisfaction, and quality of life. It is administered as a self report. Higher scores are indicative of better outcome. The summary scores is compiled by taking the mean of five subscales generated from the original questions. Range: Minimum score is 11.1, maximum 85.

CONTACTS AND LOCATIONS:
Overall Officials: YE TIAN, MD, PhD, Study Chair — First Affiliated Hospital of Harbin Medical University